CLINICAL TRIAL: NCT07171632
Title: Assessment of Mechanical Power Components on the Functional Lung in Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Components of Mechanical Power on the Functional Lung in ARDS
Status: Not yet recruiting | Type: Observational
Sponsor: Ramos Mejía Hospital (Other)
Collaborators: Universidad de la Republica (Other)
Responsible Party: Principal Investigator, Roberto Santa Cruz, PhD, Ramos Mejía Hospital
Other Study IDs: Escuela de Medicina, UMAG
Record Dates: First submitted 2025-08-24; First posted 2025-09-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Distress Syndrome (RDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survivors: Survivors patients > 18 years on the third day of ARDS receiving invasive mechanical ventilation (volume control mode) for at least 48 consecutive hours.
  Interventions: Other: monitoring of clinical and ventilatory variables

INTERVENTIONS:
Other: monitoring of clinical and ventilatory variables — Monitoring clinical data

SUMMARY:
Mechanical power (MP) is a composite variable that integrates static and dynamic respiratory parameters and has been associated with ventilator-induced lung injury (VILI). MP is predominantly delivered to the reduced functional lung size, commonly referred to as the "baby lung" (BL). Functional lung size, in turn, is closely related to respiratory system compliance (Crs). Previous studies have demonstrated an association between MP normalized to compliance (MP/Crs) and mortality. Moreover, evidence suggests that VILI associated with MP/Crs results primarily from the combined effect of its components rather than from any single component in isolation.

The objective of this study is to evaluate both the overall and the relative contribution of each component of mechanical power, normalized to compliance (MP/Crs), to in-hospital mortality in patients with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
In patients with acute respiratory distress syndrome (ARDS) who require mechanical ventilation (MV), each respiratory cycle transfers a quantifiable amount of mechanical energy to the lung. This energy is necessary both to expand the respiratory system and to overcome airway resistance. The total mechanical energy delivered per breath, when multiplied by the respiratory rate (RR), defines the concept of mechanical power (MP). From a pathophysiological perspective, MP is considered a key determinant of ventilator-induced lung injury (VILI), as it reflects the dynamic interaction of pressure, volume, and flow variables over time.

However, this transferred energy does not act uniformly throughout the lung. In ARDS, the functional portion of ventilated lung tissue is reduced due to edema, atelectasis, and consolidation. This remaining ventilatable lung volume is often referred to as the "baby lung" (BL). When mechanical energy is delivered to a smaller BL, the energy density (energy per unit of available tissue) increases, which may amplify local stress and strain, thereby exacerbating lung injury. Respiratory system compliance (Crs) has been widely used as a surrogate for BL size, given that lower compliance indicates a smaller proportion of functional lung available for ventilation.

Protective ventilation strategies, therefore, should aim not only to minimize the absolute amount of mechanical energy delivered but also to adapt it to the size of the BL in order to avoid excessive energy transfer and its potential for injury. For this reason, normalizing mechanical power to compliance (MP/Crs) has been proposed as a physiologically sound parameter, as it accounts for both the intensity of mechanical ventilation and the size of the lung that receives it.

Several studies have identified an association between MP/Crs and mortality in ARDS, supporting its role as a potential prognostic marker. Furthermore, emerging evidence suggests that the detrimental effect of MP/Crs on lung tissue is not explained by a single variable in isolation, but rather by the combined contribution of its components, including elastic dynamic power (related to driving pressure), resistive power (related to airflow resistance), and static elastic power (related to positive end-expiratory pressure). This highlights the need for a more granular evaluation of how each of these elements contributes to overall patient outcomes.

Therefore, to test the hypothesis that MP/Crs is independently associated with patient-centered outcomes in a well-characterized cohort of patients with ARDS, we will analyze detailed ventilatory parameters required for the calculation of mechanical power and its components. These data will be obtained from a prospectively collected cohort of intensive care unit (ICU) patients, allowing for accurate computation of MP/Crs and comprehensive evaluation of its relationship with clinically relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Diagnosis of acute respiratory distress syndrome
* Receiving invasive mechanical ventilation (volume control mode) for at least 48 consecutive hours.

Exclusion Criteria:

* Patients spontaneously breathing
* Patients under non-invasive support therapies
* Patients receiving ventilation through a tracheostomy cannula at any time during the first 48 h
* Patients that receiving pressure-controlled ventilation or any modality other than volume-controlled
* Patients with missing data for calculating mechanical power (MP).
* Patients with chronic pulmonary disease
* Patients with a high risk of death within 3 months for reasons other than ARDS
* Patients having made the decision to withhold life-sustaining treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years with acute respiratory distress syndrome receiving invasive mechanical ventilation for at least 48 consecutive hours
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
Mechanical Power normalized to compliance (MP/Crs) and in-hospital mortality | MP/Crs: day 3. Mortality: from enrollment until hospital discharge.
  Mechanical Power (MP) will be calculated using ventilator-derived parameters (tidal volume in mL, driving pressure in cmH₂O, inspiratory flow in L/s, and respiratory rate in breaths/min). This value will then be normalized to respiratory system compliance (Crs, in mL/cmH₂O) to obtain MP/Crs. The reported outcome will be a single aggregated measure, expressed in Joules per minute cmH2O (J/min/cmH2O), assessed on the third day of mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Angulo, PhD, Study Chair — Hospital de Clínicas "Dr. Manuel Quintela" Faculty of Medicine, Universidad de la República (Udelar) Montevideo, Uruguay; Antonella Gómez, MD, Study Director — Hospital de Clínicas "Dr. Manuel Quintela" Faculty of Medicine, Universidad de la República (Udelar) Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Santa Cruz R, Nadur J, Jara M, Navarrete M, Gagliardi J, Esquinas A, Marini JJ. Should Mechanical Power Be Normalized to Compliance? Respir Care. 2025 Jul 23. doi: 10.1177/19433654251360618. Online ahead of print. No abstract available. PMID 40711841
- [Background] Vassalli F, Pasticci I, Romitti F, Duscio E, Assmann DJ, Grunhagen H, Vasques F, Bonifazi M, Busana M, Macri MM, Giosa L, Reupke V, Herrmann P, Hahn G, Leopardi O, Moerer O, Quintel M, Marini JJ, Gattinoni L. Does Iso-mechanical Power Lead to Iso-lung Damage?: An Experimental Study in a Porcine Model. Anesthesiology. 2020 May;132(5):1126-1137. doi: 10.1097/ALN.0000000000003189. PMID 32032095
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Background] Zhang Z, Zheng B, Liu N, Ge H, Hong Y. Mechanical power normalized to predicted body weight as a predictor of mortality in patients with acute respiratory distress syndrome. Intensive Care Med. 2019 Jun;45(6):856-864. doi: 10.1007/s00134-019-05627-9. Epub 2019 May 6. PMID 31062050
- [Background] Coppola S, Caccioppola A, Froio S, Formenti P, De Giorgis V, Galanti V, Consonni D, Chiumello D. Effect of mechanical power on intensive care mortality in ARDS patients. Crit Care. 2020 May 24;24(1):246. doi: 10.1186/s13054-020-02963-x. PMID 32448389
- [Background] Chiu LC, Lin SW, Chuang LP, Li HH, Liu PH, Tsai FC, Chang CH, Hung CY, Lee CS, Leu SW, Hu HC, Huang CC, Wu HP, Kao KC. Mechanical power during extracorporeal membrane oxygenation and hospital mortality in patients with acute respiratory distress syndrome. Crit Care. 2021 Jan 6;25(1):13. doi: 10.1186/s13054-020-03428-x. PMID 33407733
- [Background] Gattinoni L, Marini JJ, Pesenti A, Quintel M, Mancebo J, Brochard L. The "baby lung" became an adult. Intensive Care Med. 2016 May;42(5):663-673. doi: 10.1007/s00134-015-4200-8. Epub 2016 Jan 18. PMID 26781952
- [Background] Dianti J, Matelski J, Tisminetzky M, Walkey AJ, Munshi L, Del Sorbo L, Fan E, Costa EL, Hodgson CL, Brochard L, Goligher EC. Comparing the Effects of Tidal Volume, Driving Pressure, and Mechanical Power on Mortality in Trials of Lung-Protective Mechanical Ventilation. Respir Care. 2021 Feb;66(2):221-227. doi: 10.4187/respcare.07876. Epub 2020 Aug 25. PMID 32843513
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Chiumello D, Brochard L, Marini JJ, Slutsky AS, Mancebo J, Ranieri VM, Thompson BT, Papazian L, Schultz MJ, Amato M, Gattinoni L, Mercat A, Pesenti A, Talmor D, Vincent JL. Respiratory support in patients with acute respiratory distress syndrome: an expert opinion. Crit Care. 2017 Sep 12;21(1):240. doi: 10.1186/s13054-017-1820-0. PMID 28899408
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32032095/